CLINICAL TRIAL: NCT04919135
Title: Clinical Study of Mesenchymal Stem/Stromal Cell Therapy in Frailty: a Proposed Experimental Design for Therapeutic and Mechanism Investigation
Brief Title: Mesenchymal Stem/Stromal Cell Therapy in the Treatment of Frailty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VinmecISC2111
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Frailty
Keywords: Frailty; umbilical cord mesenchymal stem cells
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (UC-MSC trasnplatation) (Experimental): 1.5 x 10^6 umbilical Cord Mesenchymal Stem Cells per body kg will transplant via the intravenous at baseline, and the second transplantation will be performed 3 months after the first transplantation and combination with standard frailty treatment and supplementary medication
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells transplantation; Drug: standard frailty treatment and supplementary medication
- control arm (Other): standard frailty treatment and supplementary medication
  Interventions: Drug: standard frailty treatment and supplementary medication

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells transplantation — Patients assigned to UC-MSC administration groups will receive two administrations at a dose of 1.5 million cells/kg patient body weight via the IV route with a 3-month intervening interval
  Arms: Treatment (UC-MSC trasnplatation)
Drug: standard frailty treatment and supplementary medication — Hightamine (Hankook Korus Pharm, Korea), Total calcium (Nugale Pharmaceutical, Canada), Bioflex (Ausbiomed, Australia)

SUMMARY:
This trial is to investigate the safety and potential therapeutic efficacy of allogeneic administration of umbilical cord-derived MSCs (UC-MSCs) in combination with standard frailty treatment in Vietnam

DETAILED DESCRIPTION:
Frailty, a specific condition of increased vulnerability and reduced general health associated with aging in elderly people, is an emerging global burden requiring major implications for clinical practice and public health. The lack of standardized definition and treatment of the disease resulted in the increasing number of elders diagnosed with frailty. Recently, preclinical and clinical studies support the safety of mesenchymal stem/stromal cells (MSCs) in the treatment of frailty. However, no comprehensive study has been conducted to access the interrelationship between frailty conditions and the effects of MSC-based therapy. To fill this knowledge gap, the aim of the trial is to investigate the safety and potential therapeutic efficacy of allogeneic administration of umbilical cord-derived MSCs (UC-MSCs) in combination with standard frailty treatment in Vietnam. Moreover, this study describes the rationale, study design, methodologies, and analysis strategy currently employed in stem cell research and clinical study. This randomized case-control phase I/II trial is conducted at Vinmec Times City International Hospital, Hanoi, Vietnam between July 2021 and November 2022. In this trial, 44 patients will be enrolled and randomized into a UC-MSC administration group and control group. Both groups will receive the standard frailty treatment and supplementary medication. The UC-MSC group will receive two doses of thawed UC-MSC product at 1.5x10^6 cells/kg of patient body's weight with an intervention interval of three months. The primary outcome measures will include the incidence of prespecified administration-associated adverse events (AEs) and serious adverse events (SAEs). The potential efficacy will be evaluated based on the improvement in frailty conditions (including physical examination, patient-reported outcomes, quality of life, immune markers of frailty, metabolism analysis, and cytokine markers from patient's plasma). The clinical evaluation will be conducted at baseline and 1-, 3-, 6- and 9-months post-intervention. This clinical trial and stem cell analysis associated with patients' sampling at different timepoints seeks to identify and characterize the potential effects of UC-MSCs on the improvement of frailty based on stem cell quality, cytokines/growth factors secretion profiles of UC-MSCs, cellular senescence, and metabolic analysis of patient's CD3+ cells. The ultimate results of the study will be essential for evaluating the utility of UC-MSC therapy for the treatment of frailty and mechanism underlying these effects providing the fundamental knowledge for designing and implementing research strategy of future studies

ELIGIBILITY:
Inclusion Criteria:

* Must show signs of frailty apart from a concomitant condition as assessed by the investigator with a frailty score >=3 using the Fried Phenotype Scale.
* They showed the signs of frailty based on physician assessment, apart from a concomitant condition, by a score between 3 and 6 as denoted by the Canadian Study on Health Aging.
* Must provide written informed consent.

Exclusion Criteria:

* Score of less than or equal to 20 on the Mini-Mental State Examination (MMSE)
* Active listing (or expected future listing) for transplant of any organ.
* Clinically important abnormal screening laboratory values, including but not limited to: hemoglobin <8 g/dl, white blood cell count <3000/mm3, platelets<80,000/mm3, alkaline phosphatase > 3 times the upper limit of normal, total bilirubin > 1.5 mg/dl.
* Serious comorbid illness that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study. Including, but not limited to HIV, advanced liver or renal failure, class II/III/IV congestive heart failure, myocardial infarction, unstable angina, or cardiac revascularization within the last six months, or severe obstructive ventilator defect, COPD with GOLD D, ischemic stroke with NIHSS <5, type II diabetes with HbA1C >8.5%
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.
* Be an organ transplant recipient.
* Have a clinical history of malignancy within 5 years (i.e., patients with prior malignancy must be disease-free for 5 years), except curatively treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma if recurrence occurs.
* Have a non-pulmonary condition that limits lifespan to < 1 year.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | up to the 9-month period following treatment
  To assess safety, the number of AEs or SAEs during stem cell administration (72 h) at 1 months, 3 months, 6 months and 9 months after discharge will be evaluated

SECONDARY OUTCOMES:
Reduced activities | up to the 9-month period following treatment
  Reduced activities using Community Healthy Activities Model Program for Seniors questionnaire
Slowing of mobility | up to the 9-month period following treatment
  slowing of mobility using 6-minute walk test
reduction of handgrip strength | up to the 9-month period following treatment
  reduction of handgrip strength using dynamometer
exhaustion | up to the 9-month period following treatment
  exhaustion using multidimensional fatigue inventory questionnaire
the level of pain in the knee | up to the 9-month period following treatment
  the level of pain in the knee using Western Ontario and McMaster Universities Osteoarthritis Index
respiratory function | up to the 9-month period following treatment
  respiratory function using FEV1/FVC
patients' inflammation | up to the 9-month period following treatment
  information of patients' inflammation response to umbilical cord-derived mesenchymal stem/stromal cells administration
patients' immune | up to the 9-month period following treatment
  information of patients' immune response to umbilical cord-derived mesenchymal stem/stromal cells administration
immunoregulatory properties of umbilical cord-derived mesenchymal stem/stromal cells | up to the 9-month period following treatment
  Evaluation of immunoregulatory properties of umbilical cord-derived mesenchymal stem/stromal cells
Cellular senescence | up to the 9-month period following treatment
  Measurement of cellular senescence using qPCR will be conducted in CD3+ cell population to access the expression of cyclin-dependent kinase inhibitor 2A (CDKN2A) gene, a specific biomarker indicated the cellular senescence
metabolic profiles of CD3+ cells | up to the 9-month period following treatment
  metabolic profiles of CD3+ cells via Seahorse XF Cell Mito Stress Test Kit and Seahorse XF Cell Glycolysis Stress Test Kit (Agilent Technologies)

CONTACTS AND LOCATIONS:
Overall Officials: Liem Thanh Thanh, Prof, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tompkins BA, DiFede DL, Khan A, Landin AM, Schulman IH, Pujol MV, Heldman AW, Miki R, Goldschmidt-Clermont PJ, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Da Fonseca M, Golpanian S, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Green G, Oliva AA, Hare JM. Allogeneic Mesenchymal Stem Cells Ameliorate Aging Frailty: A Phase II Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1513-1522. doi: 10.1093/gerona/glx137. PMID 28977399
- [Background] Golpanian S, DiFede DL, Pujol MV, Lowery MH, Levis-Dusseau S, Goldstein BJ, Schulman IH, Longsomboon B, Wolf A, Khan A, Heldman AW, Goldschmidt-Clermont PJ, Hare JM. Rationale and design of the allogeneiC human mesenchymal stem cells (hMSC) in patients with aging fRAilTy via intravenoUS delivery (CRATUS) study: A phase I/II, randomized, blinded and placebo controlled trial to evaluate the safety and potential efficacy of allogeneic human mesenchymal stem cell infusion in patients with aging frailty. Oncotarget. 2016 Mar 15;7(11):11899-912. doi: 10.18632/oncotarget.7727. PMID 26933813
- [Derived] Hoang VT, Le DS, Hoang DM, Phan TTK, Ngo LAT, Nguyen TK, Bui VA, Nguyen Thanh L. Impact of tissue factor expression and administration routes on thrombosis development induced by mesenchymal stem/stromal cell infusions: re-evaluating the dogma. Stem Cell Res Ther. 2024 Feb 27;15(1):56. doi: 10.1186/s13287-023-03582-3. PMID 38414067
- [Derived] Hoang DM, Nguyen KT, Hoang VT, Dao LTM, Bui HT, Ho TTK, Nguyen TTP, Ngo ATL, Nguyen HK, Thanh LN. Clinical Study of Mesenchymal Stem/Stromal Cell Therapy for the Treatment of Frailty: A Proposed Experimental Design for Therapeutic and Mechanistic Investigation. J Gerontol A Biol Sci Med Sci. 2022 Jul 5;77(7):1287-1291. doi: 10.1093/gerona/glab326. PMID 34718548